CLINICAL TRIAL: NCT07223255
Title: Gastrointestinal Response of Pediatric Cystic Fibrosis Patients on Mediterranean Diet
Acronym: MedDiet CF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Julie.L.Sanville, Assistant Professor of Pediatrics, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 02003100; P30DK117469 (NIH)
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis (CF); Cystic Fibrosis Gastrointestinal Disease
Keywords: cfmed; meddiet; meddiet cf; mediterannean diet; cystic fibrosis; CF with Mediterranean diet
MeSH Terms: conditions — Cystic Fibrosis | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- med diet (Experimental): Mediterranean diet
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: Mediterranean diet — Patients enrolled in this study will follow a Mediterranean diet for a 6 month period.

SUMMARY:
There is no study to date that has evaluated the impact or effect of a Mediterranean diet in children with CF. The goal of this study would be to help provide better guidance around questions we, as CF care providers continue to receive from patients and families about how to best promote overall health in pediatric cystic fibrosis from a dietary perspective. Currently, the updated nutritional recommendations are variable and broad. Parents continue to search for more concrete guidance about how best to promote long-term health given the ever-increasing life expectancy of cystic fibrosis patients in this new area of advanced therapeutics. Given the changing landscape of the CF care in general, children are less likely to struggle with early life malnutrition, and it is becoming increasingly clear that high fat, high calorie diets are not beneficial nor are necessary for all children with CF.

DETAILED DESCRIPTION:
The dietary needs of children with Cystic Fibrosis continue to change. With the advent of highly effective modulator therapy, these needs are profoundly shifting away from the standard advice of high calorie, high fat to varied, regular and moderated calorie. Obesity is a problem we now confront with regularity and has prompted the need for more specific, dietary advice to parents who are eager to find sustainable meal plans that promote health overall.

There is significant data to suggest that the Mediterranean Diet is the pinnacle of dietary health in everything from metabolic syndrome to ADHD in children. As we look to shift away from the standard approach, we are left to consider how specific dietary intervention may be able to support children with cystic fibrosis. Recent studies suggest Mediterranean diet and those similar were associated with increased abundance of fiber degrading bacteria like Ruminococcus as well as subclinical decreases in fecal calprotectin, a marker of gastrointestinal inflammation. In other inflammatory disease, the Mediterranean diet has also been considered as an adjunctive therapy in mild Crohn's and well as ulcerative colitis disease given its anti-inflammatory properties. Specifically in UC, notable microbiome shifts toward increased production of short chain fatty acids which can have a protective, immunomodulatory role in the gut. Data has shown that the CF gut microbiome is different than it's healthy counterparts and often described as a mix of dysbiosis and low grade chronic inflammation. If we could address the underlying inflammation and dysbiosis in a substantial way with an anti-inflammatory dietary intervention, there is potential to decrease the burden of GI disease and symptomatology that persists despite the widespread use of highly effective modulator therapy.

AIM 1: To test the hypothesis that adherence to a Mediterranean Diet will result in alterations to the gastrointestinal microbiome. We would plan to collect fecal samples for microbiota sequencing before starting a strict Mediterranean diet and then again after completion to assess for specific alterations or signatures in microbial diversity as well as other cytokine or metabolomic alterations. Our translational research core already has infrastructure set up for this process through the Dartmouth Infant and Child CF Cohort Study and many of our families are already familiar with this process.

AIM 2: To test the hypothesis that adherence to a Mediterranean Diet will result in reduction in subclinical markers of gastrointestinal inflammation. Stool calprotectin measurements from samples before and after the study period will allow us to assess for alterations.

AIM 3: To test the hypothesis that adherence to a Mediterranean Diet will result in improvement in gastrointestinal symptoms, we would also employ the PAGY-SYM, which is a widely used gastrointestinal symptom tracker to identify any significant changes in GI symptomatology before and after the anticipated diet window.

AIM 4: To test the hypothesis that adherence to a Mediterranean Diet will result in normalization of anthropometric data we will collect clinical information on subject weight, height, BMI Z score as well as mid upper arm circumference as a way to measure relative nutritional status and fat storage.

Study Endpoints:

Primary: Subjects will adhere to 6 months of exclusive Mediterranean Diet and have post diet intervention analysis of 16s and metagenomic sequencing, cytokine and metabolomic analysis for microbiome assessment.

Secondary: Fecal calprotectin as a marker of intestinal inflammation. Patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) for symptom reporting.

ELIGIBILITY:
Inclusion Criteria:

* Male and female pediatric patient with cystic fibrosis age 3 and older
* Nutritional status defined as a BMI Z-score of at least -1 or above
* Confirm diagnosis of CF defined by 2 CF causing mutations on genetic testing or sweat chloride greater than 60 mEq/L
* Children with pancreatic insufficient CF and on PERT
* Children with pancreatic sufficient CF not on PERT
* Child must be on a full, solids based diet
* Family willing to child adhere to an exclusive Mediterranean style diet for a period of 6 months
* Child must be able to follow-up at regular CF clinic visits and attend any additional study visits if necessary

Exclusion Criteria:

* Children with malnutrition
* Children who require nutritional supplementation via any type of feeding tube
* Children with poorly controlled CF lung disease
* Children with advanced CF liver disease
* Children with a comorbid gastrointestinal disease such as celiac disease, Crohn's disease or other malabsorptive process to be reviewed by PI
* Children with significant food allergies or other gastrointestinal allergy
* Family is unwilling to adhere to prescribed dietary intervention

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Metagenomic sequencing | 6 months
  Subjects will adhere to 6 months of exclusive Mediterranean Diet and have post diet intervention analysis of 16s and metagenomic sequencing, cytokine and metabolomic analysis for microbiome assessment.

SECONDARY OUTCOMES:
Fecal calprotectin | 6 months
  Fecal calprotectin as a marker of intestinal inflammation. Patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) for symptom reporting.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dartmouth Health Children's, Manchester, New Hampshire

IPD SHARING:
Plan to Share IPD: No